CLINICAL TRIAL: NCT02362867
Title: Balanced Knee System Clinical Protocol for IRB Approval
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ortho Development Corporation (Industry)
Collaborators: St. Mark's Hospital (Unknown); Salt Lake Orthopaedic Clinic (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R-07-0017
Record Dates: First submitted 2015-02-09; First posted 2015-02-13 (Estimated); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Osteoarthritis, Knee; Rheumatoid Arthritis of Knee; Post-traumatic Osteoarthritis of Knee Nos; Valgus Deformity
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Total Knee Replacement (No Intervention): Total knee replacement is indicated for patients suffering from severe knee pain and disability. Specific indications include femoral, tibial and patellar replacement due to degenerative bone disease such as osteoarthritis, rheumatoid arthritis, primary and secondary traumatic arthritis, polyarthritis, collagen disorders, avascular necrosis of the femoral condyles, or complications from a previous prosthesis. The Balanced Knee System (BKS) will be used to treat patients undergoing a total knee replacement.
  Interventions: Device: Balanced Knee System

INTERVENTIONS:
Device: Balanced Knee System — A multi-compartmental total knee replacement providing a system of components for primary posterior cruciate ligament substituting procedures. The system consists of femoral, tibial, and patellar components that allow the surgeon to select the most appropriate component combination to meet specific patient needs.
  Other Names: BKS

SUMMARY:
The protocol will define the clinical study for Ortho Development's Balanced Knee® System (BKS) for subsequent review and approval by an Institutional Review Board (IRB).This clinical study will compare the clinical outcomes of BKS to currently marketed devices.

DETAILED DESCRIPTION:
The rationale is based on the potential effectiveness of the BKS to:

* Return patient to normal activities or increase mobility by restoring knee function.
* Provide stability to enhance rehabilitation without external support.
* Eliminate or reduce knee pain.
* Assess the clinical efficacy after total knee replacement.
* Determine implant survivorship and viability.
* Evaluate patient function and satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Loss of joint configuration and joint function.
* Osteoarthritis of the knee joint.
* Rheumatoid arthritis of the knee joint.
* Post-traumatic arthritis of the knee joint.
* Moderate valgus, varus, or flexion deformities.

Exclusion Criteria:

* Any patient not experiencing a compromised quality of life by loss of joint function and/or joint configuration, or pain from arthritis disease.
* Any patient whose knee cannot be returned to normal function and normal stability through reconstructive procedures, including ligamentous balancing.
* Active infection in or near the knee joint, fever and/or local inflammation signs, and elevation of sedimentation rate unexplained by other diseases should not be treated unless preoperative infection is ruled out.
* Distant foci of infection, such as genitourinary, pulmonary, skin (chronic lesions or ulcerations), and other sites, which may result in hematogenous spread to the implant site.
* Rapid joint destruction or bone absorption apparent on roentgenograms.
* Neuromuscular disorders in which the potentially adverse effects on prosthesis function are not outweighed by the benefits gained by the patient from usage of the prosthesis.
* Mental disorders which would compromise essential patient post-operative care.
* A painless, stable arthrodesis in a functional position.
* Allergic reactions to implant materials, and/or tissue reactions to the products of corrosion or wear.
* Skeletal immaturity.
* Any patient who is unwilling or unable to comply with post-operative instructions or clinical study requirements.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2003-01 (Actual); Primary Completion 2019-06-02 (Actual); Study Completion 2019-06-02 (Actual)

PRIMARY OUTCOMES:
Evaluate effectiveness of the BKS by assessing complications during surgery and the post-operative follow-up period | 1-10 years

SECONDARY OUTCOMES:
Assess the effectiveness of the BKS by analyzing radiographic evidence and clinical data. | 1-10 years
Identify any surveillance issues regarding the device design and surgical approach used refinement of the surgical technique | 1-10 years
Evaluate device performance through the use of the Knee Society Score, Short Form-36 Health Survey, and radiographic evaluation. | 1-10 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael H. Bourne, M.D., Principal Investigator — Salt Lake Orthopaedic Clinic